CLINICAL TRIAL: NCT06137183
Title: A Phase II, Multicenter Induction Study With an Active Treatment Extension to Evaluate the Efficacy, Safety, and Pharmacokinetics of Vixarelimab in Patients With Moderate to Severe Ulcerative Colitis
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Vixarelimab in Participants With Moderate to Severe Ulcerative Colitis (UC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on a futility analysis, which suggested that the Moonglow study was unlikely to meet its primary endpoint.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GA44839; 2023-506655-19-00 (EU CTIS Number)
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Ulcerative Colitis
Keywords: Inflammatory Bowel Disease; Gastrointestinal Disease; Ulcerative Colitis; Colitis
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases; Gastrointestinal Diseases; Colitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vixarelimab Dose Regimen 1 (Experimental): Participants will receive vixarelimab subcutaneously (SC) during the induction period and the optional ATE period.
  Interventions: Drug: Vixarelimab
- Vixarelimab Dose Regimen 2 (Experimental): Participants will receive vixarelimab SC during the induction period and the optional ATE period.
  Interventions: Drug: Vixarelimab
- Placebo (Placebo Comparator): Participants will receive placebo SC during the induction period and vixarelimab SC during the optional ATE period.
  Interventions: Drug: Vixarelimab; Drug: Placebo

INTERVENTIONS:
Drug: Vixarelimab — Vixarelimab will be administered as per the schedule specified in the respective arms.
  Other Names: RO7622888; KPL-716
Drug: Placebo — Vixarelimab matching placebo will be administered as per the schedule specified in the respective arms.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics (PK) of vixarelimab compared with placebo in participants with moderate to severe UC who have demonstrated inadequate response to, loss of response to, or intolerance to prior conventional or advanced therapy.

DETAILED DESCRIPTION:
This study consists of two periods:

1. An induction period which will test the induction of clinical remission;
2. An optional active treatment extension (ATE) period which will explore durability of clinical response and remission in which all participants will receive vixarelimab.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UC for at least 3 months
* Moderately to severely active UC, assessed by mMS
* Inadequate response, loss of response to, or intolerance to conventional or advanced therapies for UC

Exclusion Criteria:

* Diagnosis of Crohn's disease or indeterminate colitis
* Suspicion of ischemic, radiation, microscopic, or infectious colitis
* Prior colectomy
* Inadequate response or loss of response to previous treatment of UC with tofacitinib, upadacitinib, or other systemic janus kinase (JAK) inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants With Clinical Remission | Week 12
  Clinical remission is defined as the Modified Mayo Score (mMS) of ≤ 2, including stool frequency subscore of ≤ 1, rectal bleeding subscore of 0, and endoscopy subscore of ≤ 1. The mMS is a composite of stool frequency, rectal bleeding, and endoscopy with each component having a scoring range of 0-3. The mMS has a total score range of 0-9 with higher scores indicating greater disease severity.

SECONDARY OUTCOMES:
Proportion of Participants With Clinical Response | Week 12
  Clinical response is defined as decrease from baseline in the mMS by ≥2 and ≥ 30% reduction from baseline, with either a decrease of ≥1 in the rectal bleeding subscore or an absolute rectal bleeding subscore of ≤1. The mMS is a composite of stool frequency, rectal bleeding, and endoscopy with each component having a scoring range of 0-3. The mMS has a total score range of 0-9 with higher scores indicating greater disease severity.
Proportion of Participants With Endoscopic Improvement | Week 12
  Endoscopic improvement is defined as a mayo endoscopy subscore of ≤ 1. Mayo endoscopy subscore has a score range of 0 (normal appearance of mucosa) to 3 (severe disease).
Proportion of Participants With Endoscopic Remission | Week 12
  Endoscopic remission is defined as a mayo endoscopy subscore of 0. Mayo endoscopy subscore has a score range of 0 (normal appearance of mucosa) to 3 (severe disease).
Number of Participants With Adverse Events (AEs) by Severity | Up to Week 56
  The AEs will be graded according to the Division of AIDS (DAIDS) table for grading the severity. The toxicity level is graded from grade 1 (lowest toxicity) to 4 (highest toxicity).
Serum Concentration of Vixarelimab | Up to Week 56
Proportion of Participants With Anti-drug Antibodies (ADAs) to Vixarelimab | Up to Week 56

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial, Study Director — Genentech, Inc.
Locations (122):
- United States (20):
  - Gulf Coast Gatroenterology, Fairhope, Alabama
  - OM Research LLC - Camarillo - ClinEdge - PPDS, Camarillo, California
  - UCLA Clinical and Translational Research Center, Los Angeles, California
  - Facey Medical Foundation - Mission Hills, Mission Hills, California
  - Clinical Applications Laboratories, Inc., San Diego, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Regenerate Primary Medical, Miami, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida
  - Orlando Gastroenterology, P.A., Orlando, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Henry Ford Health System, Novi, Michigan
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - Delta Gastroenterology & Endoscopy Center, Southaven, Mississippi
  - Strong Memorial Hospital, Rochester, New York
  - Carolina Digestive Diseases, Greenville, North Carolina
  - Ohio Gastroenterology and Liver Institute, Cincinnati, Ohio
  - North Shore Gastroenterology, Westlake, Ohio
  - Tyler Research Institute, LLC, Tyler, Texas
  - University of Utah - Health Sciences Center - PPDS, Salt Lake City, Utah
- Belgium (2):
  - CHU St Pierre (St Pierre), Brussels
  - UZ Leuven, Leuven
- Brazil (12):
  - Cliagen Clinica de Atençao em Gastroenterologia, Especialidades e Nutriçao, Salvador, Estado de Bahia
  - L2 Ip - Instituto de Pesquisas Clinicas Ltda - ME, Brasília, Federal District
  - Centro Digestivo de Curitiba, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre HCPA PPDS, Pôrto Alegre, Pará
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas da Faculdade de Medicina de Botucatu (HCFMB), Botucatu, São Paulo
  - Centro de Estudos Clinicos do Interior Paulista, Jaú, São Paulo
  - Pesquisare Saude, Santo André, São Paulo
  - Praxis Pesquisa Médica, Santo André, São Paulo
  - Kaiser Hospital Dia, São José do Rio Preto, São Paulo
  - Hospital Sirio-Libanes, São Paulo, São Paulo
  - Hospital Universitario Clementino Fraga Filho - UFRJ, Rio de Janeiro
- China (15):
  - West China Hospital - Sichuan University, Chengdu
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - Qilu Hospital of Shandong University, Jinan
  - Jinhua municipal central hospital, Jinhua
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The First Affiliated Hospital of Ningbo University(Ningbo First Hospital), Ningbo
  - Shengjing Hospital of China Medical University, Shenyang
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Wuxi People's Hospital, Wuxi
  - General Hospital of Ningxia Medical University, Yinchuan
- Czechia (4):
  - SurGal Clinic s.r.o., Brno
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - PreventaMed s.r.o., Olomouc
  - Endohope klinika s. r.o., Prague
- France (4):
  - CHU Nice - Hopital de l'Archet 2, Nice
  - Hospices Civils de Lyon Centre hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Saint-Etienne - Hopital Nord, Saint-Etienne
  - CHU de Nancy-Hopital Brabois Adulte, Vandœuvre-lès-Nancy
- Germany (4):
  - Charite - Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Halle (Saale), Halle
  - Universitatsklinikum Schleswig-Holstein - Kiel, Kiel
  - Universitaetsklinikum Ulm, Ulm
- Greece (6):
  - Evangelismos General Hospital of Athens, Athens, Attica
  - Sotiria General Hospital of Athens, Athens
  - Alexandra Hospital, Athens
  - University General Hospital of Heraklion, Heraklion
  - Iatriko Palaiou Falirou, Palaió Fáliro
  - Tzaneio General Hospital, Piraeus
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Meir Medical Center, Kfar Saba
  - Sheba Medical Center - PPDS, Ramat Gan
- Italy (8):
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi-Via Massarenti, Bologna, Emilia-Romagna
  - Fondazione Policlinico Universitario A Gemelli-Rome, Rome, Lazio
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Turin, Piedmont
  - Azienda Ospedaliero - Universitaria di Cagliari, Monserrato, Sardinia
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello, Palermo, Sicily
  - IRCCS Ospedale Sacro Cuore Don Calabria, Negrar, Veneto
- Mexico (4):
  - Hospital Puerta de Hierro Sur, Tlajomulco de Zúñiga, Jalisco
  - Accelerium, S. de R.L. de C.V. - PPDS, Monterrey, Nuevo León
  - Medical Care & Research SA de CV, Mérida, Yucatán
  - Hospital Angeles Chihuahua, Chihuahua City
- Poland (18):
  - Melita Medical Sp. Z O. O., Wroclaw, Lower Silesian Voivodeship
  - EuroMediCare Szpital Specjalistyczny z Przychodni? we Wroc?awiu, Wroclaw, Lower Silesian Voivodeship
  - Clinical Trials UMED Sp. z o. o., ?ód?
  - Szpital Zakonu Bonifratrow Sw. Jana Bozego w Lodzi sp. z o.o., ?ód?
  - Medical Center Kermed, Bydgoszcz
  - Polimedica PTG Kielce, Kielce
  - MZ Badania Slowik Zymla Sp.j., Knurów
  - Topolowa Medicenter Mrozek & Wspolnicy Spolka Jawna, Krakow
  - Allmedica Badania Kliniczne sp. z o.o. sp.k., Nowy Targ
  - Office of Jaroslaw Kierkus, Dr n Med, Otwock
  - Endoskopia Sp. z o.o., Sopot
  - Sonomed Sp. z o.o., Szczecin
  - Centrum Medyczne UNO-MED-Tarnow, Tarnów
  - NZOZ FORMED sp zo.o., Wadowice
  - Centrum Zdrowia MDM, Warsaw
  - Niepubliczny Zaklad Opieki Zdrowotnej VIVAMED, Warsaw
  - PlanetMed, Wroc?aw
  - Przychodnia VISTAMED, Wroc?aw
- Serbia (6):
  - Clinical Hospital Center Dragisa Misovic Dedinje, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Beograd-zemun
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Centre of Vojvodina, Nova Sad
  - General Hospital Djordje Joanovic - Zrenjanin, Zrenjanin
- South Korea (8):
  - Inje university Haeundae Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - The Catholic University of Korea Daejeon ST. Mary?s Hospital, Daejeon
  - Yonsei University Wonju Severance Christian Hospital, Gangwon-do
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (5):
  - E-Da Hospital, Kaohsiung City
  - Chang Gung Medical Foundation, Kaohsiung Chang Gung Memorial Hospital, Niaosong Dist.
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (3):
  - The Royal London Hospital, London
  - Hammersmith Hospital, London
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing